CLINICAL TRIAL: NCT06137872
Title: The Effect of Music on Nonstress Test and Pregnant Women's Satisfaction: Randomized Controlled Study
Brief Title: The Effect of Music on Nonstress Test and Pregnant Women's Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Resmiye KAYA ODABAŞ (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor-Investigator, Resmiye KAYA ODABAŞ, Research Assistant, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KoceliU
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Music
Keywords: music; non-stress test; pregnant
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): During the non-stress test shooting, the music group was allowed to listen to music via headphones once for at least 20 minutes.
  Interventions: Other: Music Group
- Control Group (Experimental): No application was made and non-stress test shooting was performed.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Music Group — Pregnant women who came to the hospital for non-stress testing were met and informed about the study. The procedure was applied for non-stress testing. In the music group, the pregnant woman, who was assigned to the next group according to randomization during the non-stress test, was allowed to listen to music with disposable headphones for at least 20 minutes until the procedure was completed. At the same time, the mother will be asked to close her eyes and be relaxed. Headphones used to prevent infection were given to the pregnant woman as a gift at the end of the procedure.
  Arms: Music Group
Other: Control Group — Pregnant women who came to the hospital for non-stress testing were met and informed about the study. The procedure was applied for non-stress testing. During the non-stress test, routine non-stress test was performed on the pregnant control group, which was assigned to the next group according to randomization.
  Arms: Control Group

SUMMARY:
This study was conducted as a randomized controlled trial. This study was conducted to determine the effect of music on nonstress test and pregnant woman's satisfaction. The study was conducted with pregnant women who applied for non-stress testing at a hospital in Samsun, Turkey, between September 2021 and September 2022. Pregnant women who met the research criteria were divided into two groups: physical and control groups. The research was completed experimentally with a total of 111 pregnant women, 56 experimental and 55 control. The researcher had a face-to-face interview with all the pregnant women and filled out the "Pregnant Introduction Form". Then, the vital signs of the pregnant women were taken and the pregnant women were placed in the left side-lying position. Fundus height, situs and position were determined using Leopold maneuvers. During the non-stress test shooting, the music group was allowed to listen to music for at least 20 minutes during the NST period. No intervention was made to the control group. After the non-stress test is completed, the "Satisfaction Evaluation Scale" is taken by the pregnant woman herself. The "Nonstress Test Monitoring Form" was filled out by the researcher through notification. The data of the study were evaluated using the Statistical Package for the Social Sciences program. All data were first analyzed by Kolmogorov-Smirnov for conformity with normal distribution. were evaluated and then analyzed according to their suitability for normal distribution. For descriptive statistics, percentage across the board, arithmetic mean±standard deviation for those with normal distribution, median and minimum-maximum values for those that did not fit were used. In the analysis of the data, student t test and ANOVA test were used for those that were suitable for normal distribution, and Mann-Whitney U and Kruskal Wallis tests were used for those that were not suitable for normal distribution. Type 1 error level was taken as 0.05.

DETAILED DESCRIPTION:
Aim: To determine the effect of music on non-stress test and pregnant woman's satisfaction.

Hypotheses:

H01: There is a difference between the non-stress test results of pregnant women who received music and the control group pregnant women.

H02: There is no difference between the satisfaction levels of pregnant women who received music and the control group pregnant women.

Method: The research was conducted in the non-stress test room in the gynecology outpatient clinic of a hospital in Samsun. The population of the research consisted of pregnant women who applied to the non-stress test room for non-stress test examination after having a pregnancy follow-up at the gynecology outpatient clinic of this hospital.

Sample Size: The sample number of the study was calculated according to the power analysis performed with the G Power 3.1.9.2 program. Accordingly, for the use of t-test in independent groups, effect size: 0.5, alpha = 0.05 and power: 0.80 were calculated and a total of at least 51 pregnant women were included in each group. 102 pregnant women were calculated. In order to increase the analysis power of the research, the sample size was completed with 111 pregnant women (music group: 56, control group: 55). The pregnant women in the music group and the control group were stratified according to age and the groups were distributed homogeneously.

provided. Which group the participants would be in was determined by full randomization technique on the website www.randomizer.org.

Data Collection Tools The data of the study were collected with the Pregnant Introduction Form, non-stress Monitoring Form and Satisfaction Evaluation Scale created by the researcher.

Pregnant Introduction Form: This form was developed by the researcher. It consists of questions including socio-demographic and obstetric characteristics and vital signs of pregnant women.

Nonstress Test Monitoring Form: This form was developed by the researcher and is the form preferred by pregnant women during non-stress examination.

It consists of questions about the music genre, thoughts about non-stress, and findings about non-stress for the researcher to evaluate the non-stress result. It consists of a total of 15 questions that determine pregnant women's thoughts about non-stress and include findings regarding non-stress. Non-stress results of the pregnant women were evaluated by the researcher. If there was any doubt in the evaluation, it was re-evaluated with the gynecologist.

Reactive non-stress; It was defined as the presence of at least two fetal movements within a 20-minute period, parallel to the movements, accelerations in the fetal heart rate that were more than 15 beats above the basal heart rate and lasted more than 15 seconds.

Nonreactive non-stress; It was defined as the absence of fetal movements or the presence of fetal movements, but accelerations of less than 15 beats and lasting less than 15 seconds within a 20-minute period.

Satisfaction Evaluation Scale: This scale was adapted by researchers similar to the "Visual Analog Scale (VAS)" usage principles. One end of VAS is "very good" and the other end is "very bad".

It is a scale that is evaluated by individuals by making markings on a horizontal or vertical line of 10 cm or 100 mm. This line may be just a straight line, or it may be divided at equal intervals or have descriptive words placed on the line. VAS is used to make some values that cannot be measured numerically measurable. In this scale, in order to evaluate whether the pregnant women in the music group were satisfied with the music during the non-stress shooting, the numbers between 0 and 10 were placed on a vertical line, where they would indicate with a cross (X) the point corresponding to their satisfaction with the procedure as a result of the application. In the scale, 0 points indicate "I was not satisfied at all" with the application result, and 10 points indicate "I was very satisfied" with the application result.

Collection of Data After obtaining the necessary ethics committee and institutional permission to conduct the study, the institution was visited and the pregnant women who came for non-stress examination were met. Pregnant women who meet the research criteria during working hours An explanation will be made about the purpose of the research, its content and the methods to be applied, and those who want to participate in the study are determined. Then, a random number generation program determines which group the pregnant women will be in.

They were divided into two groups: music and control groups using the "Research Randomizer". Thus, each pregnant woman's number and group number were determined and recorded. Oral and written consent of those who accepted the research Their consent was taken. The researcher had a face-to-face interview with all the pregnant women and filled out the "Pregnant Introduction Form". Then, the vital signs of the pregnant women will be taken and the pregnant women will be placed in the left side-lying position.

Fundus height, situs and position were determined using Leopold maneuvers. During the NST shooting, the music group was allowed to listen to music for at least 20 minutes during the non-stress. In the control group, no intervention was given.

It will not be done. After the nonstress test was completed, the "Satisfaction Evaluation Scale" was filled out by the pregnant woman through self-report, and the "Nonstress Test Follow-up Form" was filled out by the researcher. The interview number specified in the survey form will be written in the upper right corner of the Nonstress Test paper, and a copy of the nonstress test paper was taken with the Adobe Scan scanner installed on the smartphone device.

Statistical analysis The data of the study were evaluated using the Statistical Package for the Social Sciences (SPSS) program. All data were first evaluated with Kolmogorov-Smirnov for suitability for normal distribution, and then analyzed according to their suitability for normal distribution. For descriptive statistics, percentage across the board, arithmetic mean±standard deviation for those with normal distribution, median and minimum-maximum values for those that did not fit were used. In the analysis of the data, student t test and ANOVA test were used for those suitable for normal distribution, Mann-Whitney U and Kruskal test for those not suitable for normal distribution.

Wallis test was used. Type 1 error level was taken as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for Inclusion of Volunteers in the Research:
* Are between the ages of 18-35,
* Pregnancy week 32 and above,
* Having a singleton and live pregnancy,
* Have had non-stress test at least once before,
* Able to speak and understand Turkish,
* Pregnant women who were at least primary school graduates were included in the study.

Conditions to be met before Nonstress Testing

* Eating at least two hours before the non-stress test,
* Do not smoke, drink alcohol or use drugs for at least two hours before the non-stress test,
* Do not engage in vigorous activity for at least two hours before the non-stress test,
* Nonstress urinates just before the test,
* Basal heart rate is 110-160 beats per minute

Exclusion Criteria:

* Criteria for Excluding Preganat in the Research
* Having uterine contraction as a result of nonstress test,
* In any situation that develops acutely during the non-stress test,
* Those who cannot complete non-stress test for any reason,
* Psychologically diagnosed (such as depression, schizophrenia)
* Having any chronic disease (such as diabetes, hypertension, heart failure)
* Having pregnancy complications (such as preeclampsia, gestational diabetes, Rh incompatibility)
* Having a history of infertility and becoming pregnant with assisted reproductive techniques,
* Having a problem identified in the fetus (anomaly, intrauterine growth retardation and cardiovascular disease),
* Pregnant women who provided incorrect or incomplete information were not included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Preganant
Enrollment: 111 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Fetal heart rate | Immediately after non-stress test
  After the non-stress test was taken, the basal fetal heart rate on the non-stress test paper was calculated.
Variability | Immediately after non-stress test
  After the non-stress test was taken, the variability rate on the non-stress test paper was calculated.
  1. Increased variability (change greater than 25 beats/min from basal heart rate)
  2. Moderate variability (6-25 beats/min change from basal heart rate)
  3. Decreased variability (3-5 beats/min change from basal heart rate)
  4. No variability (0-2 beats/min change from basal heart rate)
Presence of fetal movement | Immediately after non-stress test
  After the non-stress test was taken, the presence of fetal movement on the non-stress test paper was calculated.After the non-stress test, the presence of fetal movement will be evaluated as presence/absence on the evaluation sheet, and if there is fetal movement, the number is determined.
Presence of acceleration | Immediately after non-stress test
  After taking the non-stress test, the presence of acceleration was calculated on the non-stress test paper. After the non-stress test, the presence of acceleration was evaluated as present/absent on the evaluation sheet and, if present, the number was determined.
Time to first acceleration | Immediately after non-stress test
  As a result of the non-stress test, the time until the first acceleration was calculated.
Presence of deceleration | Immediately after non-stress test
  After taking the non-stress test, the presence of deceleration was calculated on the non-stress test paper. After the non-stress test, the presence of deceleration was evaluated as present/absent on the evaluation sheet and, if present, the number was determined.
The type of deceleration | Immediately after non-stress test
  According to the non-stress test results,
  1. Early deceleration
  2. Late deceleration
  3. Variable deceleration evaluation was performed.
Nonstress test result | Immediately after non-stress test
  Evaluations are made according to the nonstress test results
  1. Reactive (negative) non-stress test (here should be at least two fetal movements within a 20-minute period, and in parallel with the movements, the fetal heart Accelerations in which the heart rate is more than 15 beats above the basal heart rate and last more than 15 seconds It will be said to be)
  2. Nonreactive (positive) non-stress test (Absence of fetal movements or presence of fetal movements within 20 minutes It will be defined as the presence of accelerations that are less than a beat and last less than 15 seconds)
  3. Questionable non-stress test evaluation was performed.
Satisfaction Evaluation Scale | Immediately after non-stress test
  This scale was adapted by researchers similar to the "Visual Analog Scale " usage principles. Visual Analog Scale is a scale evaluated by individuals by making marks on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad". This line can be just a straight line or evenly spaced.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Sökmen, Dr, Principal Investigator — Ondokuz Mayıs University; Resmiye Kaya Odabaş, Dr, Study Chair — Kocaeli University; Bahadır Yazıcıoğlu, Dr, Study Chair — Samsun Provincial Health Directorate
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No